CLINICAL TRIAL: NCT01285401
Title: A Three Arm, Randomized, Double Blind, Placebo Controlled, Multicenter, Phase II Study to Evaluate the Efficacy of Vigantol® Oil as Add on Therapy in Subjects With Relapsing Remitting Multiple Sclerosis Receiving Treatment With 44mg Tiw of Rebif®
Brief Title: Supplementation of VigantOL® Oil Versus Placebo as Add-on in Patients With Relapsing Remitting Multiple Sclerosis Receiving Rebif® Treatment
Acronym: SOLAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR 200136-532; 2010-020328-23 (EudraCT Number)
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Rebif; VigantOL® oil; Vitamin D; Add-on treatment
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a; Single Person

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VigantOL® oil (Experimental): VigantOL oil plus Rebif in subjects with 25-hydroxy-vitamin D plasma levels below 150 nmol/L
  Interventions: Drug: VigantOL oil plus interferon beta-1a (Rebif)
- Placebo (Placebo Comparator): Placebo daily plus Rebif in subjects with 25-hydroxy-vitamin D plasma levels below 150 nmol/L
  Interventions: Drug: Placebo plus interferon beta-1a (Rebif)
- Rebif (Experimental): Rebif alone in subjects with 25-hydroxy-vitamin D plasma levels equal or higher than 150 nmol/L
  Interventions: Biological: Interferon beta-1a (Rebif®) alone

INTERVENTIONS:
Drug: VigantOL oil plus interferon beta-1a (Rebif) — VigantOL oil 6,670 International Units per day (IU/d) (167 microgram per day [mcg/day]), was administered orally for 4 weeks followed by 14,007 IU/d (350 mcg/d) administered orally for 44 weeks on top of Rebif 44mcg three times per week (tiw) administered subcutaneously.
  Arms: VigantOL® oil
Drug: Placebo plus interferon beta-1a (Rebif) — Matching placebo daily, orally administered matched placebo for 48 weeks on top of Rebif 44 mcg tiw.
  Arms: Placebo
Biological: Interferon beta-1a (Rebif®) alone — Rebif® 44 mcg tiw, sub-cutaneously alone.
  Arms: Rebif

SUMMARY:
The drug being tested is called VigantOL® oil - a very effective form of Vitamin D hormone supplement (cholecalciferol). Low levels of Vitamin D have been described to be associated with a higher risk of developing Multiple Sclerosis (MS), and it is known that up to 90% of patients with Multiple Sclerosis have Vitamin D deficiency.

Rebif® is known to be an effective treatment for slowing down the progression of MS. The purpose of this research trial is to evaluate if VigantOL® oil on top of Rebif® has any benefit on the progression of MS compared to Rebif® and placebo.

Disease activity will be assessed by clinical examination and Magnetic Resonance Imaging (MRI). The planned study treatment duration for each study participant is 48 weeks, and the study consists of a total of 8 visits. Study participants who are already passed Week 48 at the time of approval of Protocol Amendment 5 will have a study duration of 96 weeks and a total of 12 visits.

During the study, the participant will undergo physical examination, neurological assessments, safety assessments, blood tests and urinalysis (including pregnancy tests).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a relapsing-remitting form of MS
* Brain and/or spinal MRI with findings typical of MS
* A first clinical event prior to Screening.
* Disease activity
* Expanded Disability Status Scale (EDSS) score of less than, or equal to 4.0 at Screening.
* Currently treated with interferon-beta-1a 44mg (tiw) sc
* Willingness and ability to comply with the protocol
* Written informed consent

Exclusion Criteria:

* Pregnancy and lactation period
* Any disease other than MS that could better explain signs and symptoms.
* Complete transverse myelitis or bilateral optic neuritis.
* Currently receiving or use at any time of monoclonal antibodies, mitoxantrone, cytotoxic or immunosuppressive therapy (excluding systemic steroids and adrenocorticotrophic hormone [ACTH]), B cell modulating therapies (e.g. RituxiMab or BelimuMab), total lymphoid irradiation or bone marrow transplantation.
* Use of any cytokine other than interferon or anti-cytokine therapy, intravenous immunoglobulin, plasmapheresis, or any investigational drug or experimental procedure
* Use of oral or systemic corticosteroids or ACTH
* Have abnormalities of Vitamin D related hormonal system other than low dietary intake or decreased sun exposure, i.e. primary hyperparathyroidism or granulomatous disorders.
* Have an urine calcium/creatinine (mmol/mmol) ratio greater than 1.0 or hypercalcaemia
* Are taking medications that influence Vitamin D metabolism other than corticosteroids, e.g., phenytoin, barbiturates, thiazide diuretics and cardiac glycosides.
* Are taking more than 1000 IU (25 µg) of Vitamin D supplement daily.
* Have conditions with increased susceptibility to hypercalcaemia, e.g., known arrhythmia or heart disease, treatment with Digitalis, or Hydrochlorothiazide and those who suffer from nephrolithiasis.
* Have inadequate liver function
* Moderate to severe renal impairment
* Inadequate bone marrow reserve
* History or presence of serious or acute heart disease such as uncontrolled cardiac dysrhythmia or arrhythmia, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure (NYHA class 3 or 4).
* History or presence of severe depression, history of suicide attempt, or current suicidal ideation.
* Epilepsy or seizures not adequately controlled by treatment.
* Current or past alcohol or drug abuse.
* Any major medical or psychiatric illness (such as psychosis, bipolar disorder) that in the opinion of the Investigator could create undue risk to the subject or could affect adherence with the trial protocol.
* Known contra-indication to treatment with vitamin D
* Known hypersensitivity to interferon or its excipient(s)
* Known hypersensitivity to gadolinium.
* Any other condition that would prevent the subject from undergoing an MRI scan.
* Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.
* Positive HIV, hepatitis C, or hepatitis B (HBsAg and HBc antibody) serology (test performed at screening).
* Legal incapacity or limited legal capacity.
* Another current autoimmune disease, except diabetes.
* Have experienced a relapse within 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manolo Beelke, MD, PhD, Study Director — WCT Worldwide Clinical Trials GER GmbH Germany; Prof. Dr. Raymond Hupperts, MD, Principal Investigator — Dept of Neurology, Orbis Medical Center Sittard, Maastricht University, The Netherlands
Locations (38):
- Research Site, Vienna, Austria
- Denmark (5):
  - Research Site, Esbjerg
  - Research Site, Glostrup Municipality
  - Research Site, Sønderborg
  - Research Site, Vejle
  - Research Site, Viborg
- Research Site, Tallinn, Estonia
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Turku
- Germany (10):
  - Research Site, Bad Neustadt / Saale
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Erlangen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hanover
  - Research Site, Münster
  - Research Site, Regensburg
  - Research Site, Rostock
- Research Site, Cefalù, Italy
- Research Site, Riga, Latvia
- Research Site, Kaunas, Lithuania
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Gouda
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
  - Research Site, Sittard
- Norway (3):
  - Research Site, Bergen
  - Research Site, Lørenskog
  - Research Site, Tromsø
- Portugal (3):
  - Research Site, Amadora
  - Research Site, Lisbon
  - Research Site, Porto
- Switzerland (5):
  - Research Site, Bern
  - Research Site, Lausanne
  - Research Site, Lugano
  - Research Site, Sankt Gallen
  - Research Site, Zurich

REFERENCES:
- [Derived] Hupperts R, Smolders J, Vieth R, Holmoy T, Marhardt K, Schluep M, Killestein J, Barkhof F, Beelke M, Grimaldi LME; SOLAR Study Group. Randomized trial of daily high-dose vitamin D3 in patients with RRMS receiving subcutaneous interferon beta-1a. Neurology. 2019 Nov 12;93(20):e1906-e1916. doi: 10.1212/WNL.0000000000008445. Epub 2019 Oct 8. PMID 31594857

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 260 subject were enrolled, out of which 232 subjects were randomized and started the study. 229 subjects were treated since 3 subjects of the 232 randomized subjects were excluded from analysis as they did not received any medication.
Groups:
- VigantOL Oil Interferon Beta-1a (Rebif): Subjects with 25-hydroxyvitamin D [25(OH)D3] serum levels below 150 nano mol per liter (nmol/L) received Vigantol oil 6,670 international unit per day (IU/d) [167 microgram per day (mcg/d)] orally for 4 weeks followed by 14,007 IU/d (350 mcg/d) for 44 weeks along with of Rebif 44 mcg administered subcutaneous three times a week (tiw).
- Placebo Interferon Beta-1a (Rebif): Subjects with 25(OH)D3 serum levels below 150 nmol/L, received matching placebo for 48 weeks on top of Rebif 44 mcg administered subcutaneous tiw.
Period: Overall Study
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Started | 115 | 117
Treated | 113 | 116
Completed | 98 | 88
Not Completed | 17 | 29
Not completed — Prematurely withdrawn from the study | 17 | 29

BASELINE CHARACTERISTICS:
Population: Baseline analysis set included all randomized subjects.
Groups:
- VigantOL Oil Interferon Beta-1a (Rebif): Subjects with 25(OH)D3 serum levels below 150 nmol/L received Vigantol oil 6,670 IU/d [167 mcg/d] orally for 4 weeks followed by 14,007 IU/d (350 mcg/d) for 44 weeks along with of Rebif 44 mcg administered subcutaneous tiw.
- Total: Total of all reporting groups
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif) | Total
Number analyzed (Participants) | 115 | 117 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (8.1) | 33.6 (9.3) | 33.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 79 | 157
  Male | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Disease Activity Free Status up to Week 48
Description: Disease activity free status was defined as absence of any of the clinical and imaging parameters related to the assessment of disease activity; no relapses, no expanded disability status scale (EDSS) progression and no new gadolinium (Gd)-enhancing or relaxation time 2 (T2) magnetic resonance imaging (MRI) lesions.
Time Frame: Up to Week 48
Population: ITT set included all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
percentage of subjects | 37.2 | 35.3

2. Secondary Outcome: Percentage of Relapse-free Subjects at Week 48
Description: A relapse was defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, lasting for 24 hours and with a previous period for more than 30 days with a stable or an improving condition.
Time Frame: Week 48
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
percentage of subjects | 78.8 | 75.0

3. Secondary Outcome: Percentage of Subjects Free From Any Expanded Disability Status Scale (EDSS) Progression at Week 48
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. A confirmed EDSS progression was defined EDSS greater than or equal to 1.0 point confirmed during a visit performed 6 months later. An EDSS progression was defined as an increase of the EDSS score of at least 1.0 point compared to baseline (SD1) for subjects with a baseline EDSS ≤ 4.0. For subjects with an EDSS score of 0 at baseline (SD1), EDSS progression was defined as an increase of at least 1.5 points. A confirmed EDSS progression was defined as an EDSS progression confirmed after 24 weeks.
Time Frame: Week 48
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
percentage of subjects | 71.7 | 75.0

4. Secondary Outcome: Number od Subjects With Confirmed EDSS Progression
Description: as for outcome 3
Time Frame: Baseline upto 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
subjects | 8 | 4

5. Secondary Outcome: Cumulative Number of Relaxation Time 1 (T1) Gadolinium Enhancing Lesions at Week 48
Time Frame: 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP. Here "N" signifies number of subject analyzed for respective outcome measure.
Measure: Mean (Standard Deviation); unit: lesions per subject per scan
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 102 | 92
lesions per subject per scan | 0.36 (1.73) | 0.25 (0.67)

6. Secondary Outcome: Mean Number of Combined Unique Active (CUA) Lesions Per Subject Per Scan at Week 48
Description: CUA lesions was defined as new T1 (Gd enhancing) lesions, new Relaxation time 2 (T2) lesions, or enlarging T2 lesions.
Time Frame: 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: lesions per subject per scan
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
lesions per subject per scan | 1.09 (3.84) | 1.49 (4.31)

7. Secondary Outcome: Cumulative Number of New Combined Unique Active (CUA) Lesions at Week 48
Description: CUA lesions was defined as new T1 (Gd enhancing) lesions, new T2 lesions, or enlarging T2 lesions.
Time Frame: 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: lesions per subject per scan
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
lesions per subject per scan | 1.09 (3.84) | 1.49 (4.31)

8. Secondary Outcome: Mean Change From Baseline in the Total Volume of T2 Lesions at Week 48 (T2 Burden of Disease)
Time Frame: Baseline, 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP. Here "N" signifies number of subjects analyzed for respective outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter^3 (mm^3)
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 103 | 92
millimeter^3 (mm^3) | 130.38 (830.82) | 95.75 (401.87)

9. Secondary Outcome: Percentage of Subjects Free From T1 Gadolinium Enhancing Lesions at Week 48
Time Frame: 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
percentage of subjects | 83.2 | 70.7

10. Secondary Outcome: Percentage of Subjects Free From New T1 Hypointense Lesions (Black Holes) at Week 48
Time Frame: 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
percentage of subjects | 78.8 | 63.8

11. Secondary Outcome: Percentage of New T1 Hypointense Lesions (Black Holes) at Week 48 Within the Subgroup of New or Enlarging Non-enhancing T2 Lesions
Time Frame: 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP. Here "N" signifies number of subjects analyzed for respective outcome measure (here in the subgroup of subjects having new or enlarging T2 lesions).
Measure: Mean (Standard Deviation); unit: percentage of new T1 hypointense lesions
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 25 | 36
percentage of new T1 hypointense lesions | 20.11 (34.72) | 27.70 (39.33)

12. Secondary Outcome: Number of Subjects With Relapse
Description: Relapse was defined as neurological abnormality, either newly appearing or re-appearing, with abnormality specified by both as neurological abnormality separated by at least 30 days from onset of a preceding MS attack and Neurological abnormality lasting for at least 24 hours, absence of fever or known infection greater than 37.5 degree centigrade /99.5 degree fahrenheit , objective neurological impairment, correlating with the subject's reported symptoms, defined as either increase in at least one of the functional systems of the EDSS or increase of the total EDSS score and occurrence of paraesthesia, fatigue, mental symptoms, and/or vegetative symptoms without any additional symptom will not be classified as an MS attack.
Time Frame: Baseline upto 48 weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
subjects | 24 | 29

13. Secondary Outcome: Annualized Relapse Rate at Week 48
Description: as for outcome 12
Time Frame: 48 weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: relapse per year
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
relapse per year | 0.28 (0.59) | 0.41 (0.83)

14. Secondary Outcome: Total Number of Reported Relapses at All Time Points up to 48 Weeks
Description: as for outcome 12
Time Frame: 48 weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: number of relapse per subject
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
number of relapse per subject | 0.25 (0.53) | 0.34 (0.63)

15. Secondary Outcome: Percentage of Subjects Treated With Glucocorticoids Due to Relapses
Description: as for outcome 12
Time Frame: Baseline upto 48 weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
percentage of subjects | 15.9 | 20.7

16. Secondary Outcome: Mean Change From Baseline in the Total Volume of T1 Hypo Intense Lesions at Week 48
Time Frame: Baseline, 48 Weeks
Population: ITT analysis set consisted of all randomized subjects who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: millimeter^3 (mm^3)
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
millimeter^3 (mm^3) | 20.88 (140.56) | 18.47 (68.08)

17. Post Hoc Outcome: Percentage of Subjects With Disease Activity Free Status (Alternate Definition) at Week 48
Description: Disease activity free (DAF) status was defined as absence of any of the clinical and imaging parameters related to the assessment of disease activity; no relapses, no confirmed expanded disability status scale (EDSS) progression and no new gadolinium (Gd)-enhancing or relaxation time 2 (T2) magnetic resonance imaging (MRI) lesions. Confirmed EDSS progression was defined as an EDSS progression confirmed after 24 weeks.
Time Frame: Week 48
Population: ITT set included all randomized subjects who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of subjects
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Number analyzed (Participants) | 113 | 116
percentage of subjects | 47.8 | 37.9

ADVERSE EVENTS:
Time Frame: Baseline up to end of trial (EOT: 50 months)
Description: Safety Analysis Set: All randomized subjects who received at least 1 dose of the IMP
Arm/Group | VigantOL Oil Interferon Beta-1a (Rebif) | Placebo Interferon Beta-1a (Rebif)
Serious Adverse Events (participants affected / at risk) | 18/113 | 8/116
Other Adverse Events (participants affected / at risk) | 99/113 | 93/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VigantOL Oil Interferon Beta-1a (Rebif) (N=113) | Placebo Interferon Beta-1a (Rebif) (N=116)
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 8 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VigantOL Oil Interferon Beta-1a (Rebif) (N=113) | Placebo Interferon Beta-1a (Rebif) (N=116)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 2 | 3
Thyroid disorder (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 2
Diplopia (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 2 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 3 | 3
Glaucoma (Eye disorders) | 0 | 1
Oscillopsia (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 3 | 3
Visual impairment (Eye disorders) | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 7
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 4
Vomiting in pregnancy (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 4
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 8 | 13
Feeling cold (General disorders) | 2 | 0
Gait disturbance (General disorders) | 3 | 2
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 12 | 13
Injection site erythema (General disorders) | 4 | 0
Injection site induration (General disorders) | 0 | 1
Injection site inflammation (General disorders) | 1 | 0
Injection site irritation (General disorders) | 1 | 1
Injection site pain (General disorders) | 2 | 2
Injection site pruritus (General disorders) | 0 | 1
Injection site reaction (General disorders) | 5 | 3
Injection site swelling (General disorders) | 1 | 0
Injection site urticaria (General disorders) | 0 | 3
Irritability (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 7 | 12
Sensation of foreign body (General disorders) | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Multiple allergies (Immune system disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 4 | 2
Cystitis (Infections and infestations) | 3 | 7
Ear infection (Infections and infestations) | 2 | 1
Eye infection (Infections and infestations) | 1 | 1
Eyelid infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 1
Gastric infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 5
Gastroenteritis viral (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 1 | 0
Infected cyst (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 13 | 19
Injection site abscess (Infections and infestations) | 2 | 0
Laryngitis (Infections and infestations) | 3 | 2
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 18 | 17
Oral herpes (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pseudofolliculitis barbae (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 4 | 2
Rhinitis (Infections and infestations) | 5 | 1
Sinusitis (Infections and infestations) | 5 | 4
Skin infection (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 12 | 6
Vaginal infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 3 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Anti-thyroid antibody positive (Investigations) | 1 | 0
Antibody test positive (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Blood creatinine decreased (Investigations) | 0 | 1
Blood folate decreased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 2 | 0
Blood iron decreased (Infections and infestations) | 1 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone abnormal (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Creatine urine abnormal (Investigations) | 0 | 1
Creatinine urine increased (Investigations) | 0 | 1
Drug specific antibody present (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Thyroid function test abnormal (Investigations) | 0 | 1
Urine calcium (Investigations) | 0 | 1
Urine calcium/creatinine ratio increased (Investigations) | 1 | 0
Vitamin B12 decreased (Investigations) | 2 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Growing pains (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 5 | 4
Dystonia (Nervous system disorders) | 1 | 0
Facial neuralgia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 20 | 21
Hypoaesthesia (Nervous system disorders) | 2 | 2
Memory impairment (Nervous system disorders) | 2 | 0
Meralgia paraesthetica (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 6 | 5
Migraine with aura (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 5 | 4
Presyncope (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 3
Sciatica (Nervous system disorders) | 1 | 1
Sensory disturbance (Nervous system disorders) | 4 | 3
Syncope (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Affective disorder (Psychiatric disorders) | 0 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 5
Anxiety disorder (Psychiatric disorders) | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Delusional perception (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 2
Fear of needles (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 4
Loss of libido (Psychiatric disorders) | 0 | 1
Mood swings (Psychiatric disorders) | 2 | 0
Panic attack (Psychiatric disorders) | 0 | 3
Restlessness (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 4
Stress (Psychiatric disorders) | 2 | 0
Bladder dysfunction (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 4
Incontinence (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 4
Endodontic procedure (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 0
Mammoplasty (Surgical and medical procedures) | 1 | 0
Parotidectomy (Surgical and medical procedures) | 1 | 0
Shoulder operation (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other